CLINICAL TRIAL: NCT04383912
Title: Onabotulinum Toxin A to Improve Direct Brow Lift Outcomes
Brief Title: Onabotulinum Toxin A in Direct Brow Lift
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Ahsen Hussain, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Botox Direct Brow Lift
Record Dates: First submitted 2020-05-01; First posted 2020-05-12 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Direct Brow Lift; Scarring
Keywords: onabotulinum toxin; direct brow lift; scarring; Botox
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: This is a double masked, prospective, randomized controlled trial. Participants will function as their own internal control, with one side (i.e. brow) being randomized to the treatment arm, and the other to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computer randomization software will be used to determine whether the right or left side will receive onabotulinum toxin injection. The contralateral side will receive a placebo injection of equal volume (normal saline).
  The health care professional assisting with the procedure will not be masked to randomization. He/she will draw up the onabotulinum toxin A and placebo in two separate identical syringes marked A (right side) and B (left side). They will reference a form showing the results of the computer generated randomization, which will be kept in a study chart separate from the patient's normal oculoplastic visits. They will sign this form, as well as record the lot number of the onabotulinum toxin A and normal saline.
  The oculoplastic surgeon will visually divide each incision in half, and inject half of the volume of syringe A at each side of the right direct brow lift incision, and half of the volume of syringe B at each side of the left direct brow lift incision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- onabotulinum toxin A group (brow) (Experimental): Product name: Onabotulinum toxin A (Botox A, Allergan), 50 unit vials Product code: 93094EC
  Description: The side randomized to treatment will receive an injection of 20 units of onabotulinum toxin A as the final step of a direct brow lift surgery. The surgeon will visually divide the surgical incision in half, and divide the volume of the injection evenly between the two sides. This will be a one time administration.
  Interventions: Drug: Botox Injectable Product
- placebo group (brow) (Placebo Comparator): Product name: normal saline
  Description: The side randomized to placebo will receive an injection of normal saline as the final step of a direct brow lift surgery. The surgeon will visually divide the surgical incision in half, and divide the volume of the injection evenly between the two sides. This will be a one time administration.
  Interventions: Other: No intervention (placebo)

INTERVENTIONS:
Drug: Botox Injectable Product — The side randomized to receive treatment will be injected with onabotulinum toxin A. Wound healing, scar characteristics, and patient satisfaction will be assessed post operatively. Scarring will be assessed by the patient, medical observers and a lay observer, all masked to the treatment vs placebo side. Standardized scales will be used, and pre-operative, intra-operative, and post-operative photographs will be taken for all participants. ImageJ software will be used to analyze the photos and measure the degree of brow lift achieved on each side, to ensure this has not been affected by onabotulinum toxin injection.
  Arms: onabotulinum toxin A group (brow)
Other: No intervention (placebo) — This group (of brows) will be receiving placebo injections containing normal saline. They will be assessed in the same manner as the treatment side.
  Arms: placebo group (brow)

SUMMARY:
The brow lift is a surgical procedure that has been practiced for several decades. A typical indication is brow ptosis, which can be secondary to involutional changes or facial nerve palsies. Several techniques have been described, including direct, mid-forehead, coronal, and endoscopic approaches. Of these options, the direct brow lift allows for predictable post-operative brow contour and excellent control over the degree of lift achieved. As with any surgical procedure, with direct brow lift comes known undesirable post-operative outcomes, the most common of which is forehead paresthesia from supraorbital nerve damage. Other complications include alopecia and brow asymmetry. However, one of the main critiques of direct brow lift remains the poor cosmesis that can result from scarring just above the brow. A study conducted by Cho et al. concluded that of the main surgical techniques currently employed for treatment of brow ptosis, direct brow lifts held the highest rates of visible scarring.

Scarring can significantly impair an individuals' quality of life. This is particularly true of facial scarring, which is often difficult to conceal. Much research has been conducted in the area of treating postoperative, traumatic, and burn-related scarring. Cadet et al completed a randomized controlled trial using topical silicone gel for direct brow lift-related scarring, given the known benefit of silicone gel sheeting for the same, but did not find a significant difference between treatment and control groups. Some effective techniques described in the literature to date include long-pulsed non-ablative Nd:YAG laser, as well as intralesional steroid injection. On the rise are studies looking into the use of botulinum toxin A for treatment of unfavourable scarring and improved facial cosmesis.

Botulinum toxin is a neuromodulatory agent that has garnered usage in a variety of therapeutic and cosmetic settings. More recently, injection of botulinum toxin as a means to reduce scarring and improve outcomes in wound healing has been investigated. Several studies, including two large metaanalyses, have shown this to be an effective method of treatment. Proposed mechanisms include increased apoptosis and suppressed proliferation of fibroblasts treated with botulinum toxin, modulated via the PTEN/PI3K/Akt pathway. Park et al added to the in vitro literature by demonstrating that fibroblasts treated with botulinum toxin A produced fewer extracellular matrix proteins and pro-fibrotic factors compared to untreated cells. Another underlying mechanism that results in suboptimal wound healing is the constant contraction and relaxation of facial muscles, causing repetitive microtrauma that ultimately increases inflammation and impairs wound healing. It therefore stands to reason that by temporarily paralyzing local musculature during the post-operative period, collagen maturation can take place uninterrupted by excessive tensile forces.

Despite scarring being a widely known and undesirable complication of direct brow lift surgery, there have been no studies to date examining the use of onabotulinum toxin injection to reduce said scarring and improve outcomes. With this double masked, prospective, randomized controlled trial, the investigators aim to determine whether injection of onabotulinum toxin immediately following direct brow lift surgery can improve scores on validated patient and observer scar scales.

ELIGIBILITY:
The patient population to be studied will include patients undergoing bilateral direct brow lifts at the Victoria General Hospital in Halifax, Nova Scotia.

Patients must meet all of the following inclusion criteria, and have none of the exclusion criteria listed below.

Inclusion criteria:

* Participants must be over 18 years of age
* Participants must be able to attend outpatient appointments at the Victoria General Hospital
* Participants must be able to give informed consent

Exclusion criteria:

* Known allergy to botulinum toxin
* Previous scarring in same region of surgical procedure
* Previous botulinum toxin injection within 6 months of surgical date for direct brow lift
* Currently pregnant or breast feeding
* History of keloid or hypertrophic scarring
* History of myasthenia gravis/ neuromotor disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Effect of onabotulinum toxin A on scarring in direct brow lift surgery | 1 to 12 months
  * At 1 month following surgery, photographs will be taken of both brows. The patient will then be given a mirror, and under consistent lighting conditions and in a private setting, will complete the Patient Scar Assessment Scale (PSAS) and Visual Analog Scale (VAS), after adequate explanation of each parameter. These scores will be combined for a total score ranging from 7 to 70, again with lower numbers indicating higher patient satisfaction. A masked lay observer (consistent person with every patient) will also complete the VAS.
  * The above step will be repeated at 3 months, 6 months, and 12 months after surgery, as well as the following additional steps. Scars will be graded by a masked observer using the Observer Scar Assessment Scale (OSAS), Observer Modified Scar Assessment Scale (OMSAS), and Visual Analog Scale (VAS). These scores will be combined for a total score ranging from 11 to 81, with lower scores indicating better outcome.
Degree of brow lift achieved | Pre-operative to 12 months
  Pre-operative, intra-operative, and post-operative (at month 1, 3, 6, and 12) photographs will be taken for all participants. ImageJ software will be used to analyze the photos and measure the degree of brow lift achieved on each side, to ensure this has not been affected by botulinum toxin injection. This will be measured from the pupillary light reflex to the upper border of the eyebrow (in mm). These measurements will be done by a masked observer.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen Hussain, FRCOphth, MD, Principal Investigator — Staff surgeon (ophthalmic plastic and reconstructive surgery)
Locations (1):
- Eye Care Centre, Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Booth AJ, Murray A, Tyers AG. The direct brow lift: efficacy, complications, and patient satisfaction. Br J Ophthalmol. 2004 May;88(5):688-91. doi: 10.1136/bjo.2003.019232. PMID 15090424
- [Background] Cho MJ, Carboy JA, Rohrich RJ. Complications in Brow Lifts: A Systemic Review of Surgical and Nonsurgical Brow Rejuvenations. Plast Reconstr Surg Glob Open. 2018 Oct 15;6(10):e1943. doi: 10.1097/GOX.0000000000001943. eCollection 2018 Oct. PMID 30534495
- [Background] Price P, Tebble N. Psychological consequences of facial scarring. Chapter from Surgery in Wounds 2004, 519-526.
- [Background] Cadet N, Hardy I, Dudek D, Miszkiewicz K, Boulos P, Nguyen Q, Wong J. Prospective case-control trial evaluating silicone gel for the treatment of direct brow lift scars. Can J Ophthalmol. 2018 Feb;53(1):29-33. doi: 10.1016/j.jcjo.2017.07.017. PMID 29426436
- [Background] Tenzel PA, Patel K, Erickson BP, Shriver EM, Grunebaum LD, Alabiad CR, Lee WW, Wester ST. Split face evaluation of long-pulsed non-ablative 1,064 nm Nd:YAG laser for treatment of direct browplasty scars. Lasers Surg Med. 2016 Oct;48(8):742-747. doi: 10.1002/lsm.22543. Epub 2016 Aug 9. PMID 27505684
- [Background] Trisliana Perdanasari A, Torresetti M, Grassetti L, Nicoli F, Zhang YX, Dashti T, Di Benedetto G, Lazzeri D. Intralesional injection treatment of hypertrophic scars and keloids: a systematic review regarding outcomes. Burns Trauma. 2015 Aug 26;3:14. doi: 10.1186/s41038-015-0015-7. eCollection 2015. PMID 27574660
- [Background] Guo X, Song G, Zhang D, Jin X. Efficacy of Botulinum Toxin Type A in Improving Scar Quality and Wound Healing: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Aesthet Surg J. 2020 Apr 14;40(5):NP273-NP285. doi: 10.1093/asj/sjz165. PMID 31155638
- [Background] Yang W, Li G. The Safety and efficacy of botulinum toxin type A injection for postoperative scar prevention: A systematic review and meta-analysis. J Cosmet Dermatol. 2020 Apr;19(4):799-808. doi: 10.1111/jocd.13139. Epub 2019 Sep 12. PMID 31513335
- [Background] Zhang X, Lan D, Ning S, Jia H, Yu S. Botulinum toxin type A prevents the phenotypic transformation of fibroblasts induced by TGF-beta1 via the PTEN/PI3K/Akt signaling pathway. Int J Mol Med. 2019 Aug;44(2):661-671. doi: 10.3892/ijmm.2019.4226. Epub 2019 May 31. PMID 31173164
- [Background] Park GS, An MK, Yoon JH, Park SS, Koh SH, Mauro TM, Cho EB, Park EJ, Kim KH, Kim KJ. Botulinum toxin type A suppresses pro-fibrotic effects via the JNK signaling pathway in hypertrophic scar fibroblasts. Arch Dermatol Res. 2019 Dec;311(10):807-814. doi: 10.1007/s00403-019-01975-0. Epub 2019 Sep 9. PMID 31501922
- [Background] Shome D, Khare S, Kapoor R. An Algorithm Using Botox Injections for Facial Scar Improvement in Fitzpatrick Type IV-VI Skin. Plast Reconstr Surg Glob Open. 2018 Aug 8;6(8):e1888. doi: 10.1097/GOX.0000000000001888. eCollection 2018 Aug. PMID 30324067
- [Background] Tyers AG, Collin JRO. In: Colour atlas of ophthalmic plastic surgery. 2nd ed. Oxford: Butterworth-Heinemann, 1997, 178-82.
- [Background] Ziade M, Domergue S, Batifol D, Jreige R, Sebbane M, Goudot P, Yachouh J. Use of botulinum toxin type A to improve treatment of facial wounds: a prospective randomised study. J Plast Reconstr Aesthet Surg. 2013 Feb;66(2):209-14. doi: 10.1016/j.bjps.2012.09.012. Epub 2012 Oct 25. PMID 23102873